CLINICAL TRIAL: NCT05056701
Title: Prediction of Chronic Kidney Disease Following Pre-eclampsia: Diagnosis and Early Care
Acronym: PRECEDE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier le Mans (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CHM-2020/S8/10
Record Dates: First submitted 2021-09-16; First posted 2021-09-24 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Preeclampsia
Keywords: chronic kidney disease (CKD); preeclampsia
MeSH Terms: conditions — Pre-Eclampsia; Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- patient with preeclampsia (Experimental): Patient meeting the preeclampsia criteria or one of its complications (eclampsia, HELLP syndrome) according to the ISSHP 2018 definitions within the last 5 years
  Interventions: Other: annual follow-up during 10 years

INTERVENTIONS:
Other: annual follow-up during 10 years — an annual follow-up is carried out systematically for a total of 10 years in order to detect the subsequent occurrence of CKD

SUMMARY:
Pre-eclampsia (PE) is a pregnancy-associated syndrome of variable severity, classically defined by the combination of hypertension and proteinuria in a previously non-hypertensive or proteinuric patient. These symptoms normally resolve within 2-3 months after delivery regardless of the severity of the pre-eclampsia.

Regardless of its definition, preeclampsia is associated with an increased risk of obstetric events and, for the mother, an increased risk of developing chronic kidney disease (CKD), hypertension, diabetes and cardiovascular disease in the broad sense.

The relationship between preeclampsia and Chronic Kidney Disease is, however, complex and not fully understood.

Investigator proposes an interventional study to identify the diagnosis of Chronic Kidney Disease in patients who have developed an episode of Preeclampsia.

ELIGIBILITY:
Inclusion Criteria:

* Meeting the preeclampsia criteria or one of its complications (eclampsia, HELLP syndrome) according to the ISSHP 2018 definitions within the last 5 years
* Having signed the informed consent
* Person affiliated to social security

Exclusion Criteria:

* Patient with mental disability or language barrier preventing understanding of the study or consent
* Person deprived of liberty by judicial or administrative decision
* Person under forced psychiatric care
* Person subject to a legal protection measure

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2022-05-30 (Actual); Primary Completion 2037-05-30 (Estimated); Study Completion 2037-05-30 (Estimated)

PRIMARY OUTCOMES:
prevalence of the Chronic Kidney Disease (CKD) | until 10 years
  prevalence of the CKD is measured by the the rate of new CKD Diagnoses (according to the standard definitions)

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Chu Angers, Angers
  - Centre Hospitalier Du Mans, Le Mans

IPD SHARING:
Plan to Share IPD: No